CLINICAL TRIAL: NCT04476355
Title: Development of Physical Restraints Clinical Practice Guidelines for Critically Ill Patients and Implementation Study Using the CAN-IMPLEMENT Framework
Brief Title: Implementation of Physical Restraints Clinical Practice Guidelines for Critically Ill Patients Using the CAN-IMPLEMENT Framework
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-533
Record Dates: First submitted 2020-06-28; First posted 2020-07-20 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-06

CONDITIONS: Restraint, Physical; Intensive Care Units; Practice Guideline; Health Plan Implementation

STUDY DESIGN:
Intervention Model Description: In the same ICU, the patients in the study period were the experimental group and the former patients were the control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): In the same ICU, the former(2019-12~2020-12) patients were the control group, data collected through case system.
- experimental group (Experimental): In the same ICU, the patients in the study period were the experimental group
  Interventions: Other: Select and Tailor implementation interventions

INTERVENTIONS:
Other: Select and Tailor implementation interventions — Based on previously adapted guidelines and the assessment of innovation, adopters and practice environment for barriers and supports, the interventions mainly include patients education, practioners education and system changes.
  Arms: experimental group

SUMMARY:
Physical restraints (PR) are widely used in ICU around the world. Many institutions have suggested that the use of PR should be reduced. Clinical practice guidelines (CPGs) are a convenient way of packaging evidence and presenting recommendations to healthcare decision makers. There are currently no CPGs on PR in China, while other countries had, so we hope to be able to adapt existing guidelines to apply in Chinese context. We use the CAN-IMPLEMENT approach to adapt and implement the guidelines.

DETAILED DESCRIPTION:
Critically ill patients admitted to intensive care units (ICU) often need more invasive operations (e.g.mechanical ventilation and hemodialysis), due to the needs from their condition, which can also lead to acute pain, discomfort, sleep deprivation, agitation and delirium. Agitation, for example, can propel patients to resist the ventilator, thus increasing the oxygen consumption, causing them to accidentally remove various devices and catheters on them and even posing life-threatening risks. Therefore, the main reason for the use of physical restraints (PR) around ICU is to prevent patients from accidentally removing the catheters or devices needed to protect their safety.

Although PR was used to prevent Unplanned extubation (UE), there were many studies proved that PR is one of the risk factors that account for UE and can not protect patient safety. Indeed, its use has been proven to cause pressure injuries, worsen agitation, delirium and neurovascular complications. But PR is widely used in ICU around the world.

Many institutions have suggested that the use of PR should be reduced, for example, the Government of Ontario released the Patient Restraints Minimization Act in 2001 to "minimize the use of restraints on patients and to encourage hospitals and facilities to use alternative methods, whenever possible, when it is necessary to prevent serious bodily harm by a patient to himself or herself or to others. Registered Nurses Association of Ontario (RNAO) issued clinical practice guidelines on the alternatives to PR in February 2012, aimed to help nurses reduce the use of PR, or use it in a more reasonable and standardized way, and to provide effective alternatives of PR.

Clinical practice guidelines (CPGs) are a convenient way of packaging evidence and presenting recommendations to healthcare decision makers. But the development and updating of high-quality CPGs require substantial time, expertise and resources. Guideline adaptation is the systematic approach to the endorsement and/or modification of a guideline(s) produced in one cultural and organisational setting for application in a different context. Where high quality guidelines are already available, adaptation may be used as an alternative to de novo guideline development to customise the existing guideline to the needs of local users. There are currently no CPGs on PR in China, while other countries had, so we hope to be able to adapt existing guidelines to apply in Chinese context. We use the CAN-IMPLEMENT approach to adapt and implement the guidelines.

ELIGIBILITY:
Inclusion Criteria:

* The patient him/herself or the patient's authorized agent signed the informed consent to the study

Exclusion Criteria:

* Patients with a history of basic mental illness or cognitive impairment before admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
rate of utilization of physical restraints | 2 years
  Length of utilization of physical restraints / length of stay in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The data analyzed in this study is not included in a repository because it contains interview transcripts.